CLINICAL TRIAL: NCT05839314
Title: Effect of Huaier Granule on the Treatment of Idiopathic Membranous Nephropathy: a Multicenter, Randomized, Open-label, Parallel Controlled Study
Brief Title: Effect of Huaier Granule on the Treatment of Idiopathic Membranous Nephropathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiangmei Chen, Dr., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202009
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Nephropathy; Glomerular Diseases; Idiopathic Membranous Nephropathy
Keywords: Huaier granule; Ciclosporin; Idiopathic membranous nephropathy
MeSH Terms: conditions — Kidney Diseases; Glomerulonephritis, Membranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier group (Experimental): Patients will take Huaier granule and renin-angiotensin-aldosterone system inhibitors (RASI).
  Interventions: Drug: Huaier granule; Drug: Renin-angiotensin-aldosterone system inhibitors (RASI)
- Ciclosporin soft capsules group (Active Comparator): Patients will take Ciclosporin soft capsules and RASI.
  Interventions: Drug: Renin-angiotensin-aldosterone system inhibitors (RASI); Drug: Ciclosporin soft capsules

INTERVENTIONS:
Drug: Huaier granule — Huaier granule, oral administration, 10g each time, 3 times a day, continuous medication for 24 weeks. After 24 weeks of treatment, the dosage should be adjusted according to efficacy.
  Other Names: Jinke
  Arms: Huaier group
Drug: Renin-angiotensin-aldosterone system inhibitors (RASI) — Run-in period: All the patients should be treated with RASI for at least 4 weeks, and stop using any medicine containing Huaier or similar ingredients for at least 2 weeks before enrollment. If the patient is receiving RASI, the RASI can be continued until the end of the study. RASI can be adjusted once a week until the maximum tolerable dose based on albuminuria and blood pressure. If the patient is not receiving RASI therapy, then RASI is recommended.
  Treatment period: RASI therapy is continued throughout the trial. Check blood pressure twice daily: morning and evening.
Drug: Ciclosporin soft capsules — The initial dose of Ciclosporin soft capsules is an oral dose of 3.5mg/kg/d, divided into two equal doses, given every 12 hours. Assess the plasma concentration of CsA (valley value) every 2 weeks in the first 8 weeks. If the plasma concentration of CsA reaches 100-150ug/L, continue to maintain the dose. If the plasma concentration of CsA is below the target concentration, increase the dose of CsA. If the plasma concentration of CsA is higher than the upper limit of the target concentration, appropriate dose reduction. A single dose adjustment is 25mg/d. After increasing/decreasing the dose, CsA concentration is remeasured at intervals of 2 weeks ±3 days until the target concentration is reached.
  CsA at target concentration followed by 24 weeks of treatment, then the dosage shall be adjusted according to efficacy.
  Arms: Ciclosporin soft capsules group

SUMMARY:
This is a prospective, multicenter, randomized, open-label, parallel controlled study. The purpose of this study is to evaluate the efficacy and safety of Huaier granule on the treatment of idiopathic membranous nephropathy comparing with Ciclosporin soft capsules.

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy (IMN) is a common immune-mediated glomerular disease, accounting for 20% to 36.8% of adult nephrotic syndrome. A third of the patients will experience complete remission spontaneously, and 30%-40% of patients will develop chronic renal failure. The treatment of IMN includes supportive therapy and immunosuppressive therapy. Ciclosporin (CsA) is a kind of calcineurin inhibitor (CNI) recommended by the Kidney disease improving global outcomes (KDIGO) clinical practice guideline for IMN treatment. CsA is effective in inducing remission among patients with steroid-resistant nephrotic IMN, and studies showed the clinical remission rate was 60%-75%. However, it has a high rate of relapse during follow-up in 6-12 months.

Huaier granule is an extract from a medicinal fungus. Previous studies showed that Huaier granule reduced the excretion of proteinuria, inhibited inflammation and cellular transdifferentiation, and protect renal function.

In this study, about 30 research centers will participate. We plan to enroll 480 participants (240 cases in the experimental group and 240 cases in the control group). The planned length of patient recruitment enrolment will be 2 years and the total length of visits be 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Renal biopsy was performed before randomization and pathologically diagnosed as idiopathic membranous nephropathy;
* Anti-phospholipase a2 receptor (PLA2R) antibody is positive;
* Aged from 18 to 75, either sex;
* Tolerable doses of RASI were received for ≥4 weeks before randomization, nephrotic syndrome was not in remission and 24-hour urinary protein level was ≥3.5g/24h and < 8.0g/24h;
* The eGFR≥45ml/min/1.73m2 (Measured at least twice in 2 weeks);
* The patient is willing to sign the informed consent form.

Exclusion Criteria:

* Diagnosed as secondary membranous nephropathy;
* Rapidly progressive membranous nephropathy (eGFR decreased by 50 % compared with the baseline level within 3 months);
* Receiving renal replacement therapy;
* Diabetes and glycosylated hemoglobin (HbA1c) levels ≥ 7.0%;
* Hypertension is not well controlled (systolic blood pressure>160mmHg or diastolic blood pressure>100mmHg);
* The level of serum albumin≤20g/L;
* Resistance to treatment with CsA or other CNI, rituximab (RTX) or alkylating agents; complete remission or partial remission was obtained after treatment with CNI, RTX, or alkylating agents but there was a history of relapse within 3 months；
* Suspected infection by imaging and/or laboratory tests;
* Infectious diseases, such as hepatitis B, hepatitis C, AIDS, tuberculosis;
* History of malignant tumor;
* Hepatic dysfunction: aspartate aminotransferase (AST) concentration and alanine aminotransferase (ALT) concentration of > 1.5 × upper limit of normal;
* Allergic to Huaier granule or Ciclosporin soft capsules;
* Previous CNI treatment was ineffective;
* Complicate with any diseases that may affect efficacy and safety evaluation;
* Pregnant or lactating women, and patients (male or female) with fertility plans or unwilling to take effective contraceptive measures;
* Participating in other clinical trials or participated in other clinical studies within 3 months;
* According to the researchers, patients have diseases or conditions that increase the difficulty of enrollment or probability of loss to follow-up, such as mental illness, frequent changes in residence and work, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall clinical remission rate at 24, 48, 96 weeks | Start of randomization until 96 weeks
  Overall clinical remission rate is defined as rate of complete remission and partial remission. Complete remission is defined as a 24-h urinary protein level < 0.3g/d with normal serum albumin level and stable renal function. Partial remission is defined as 24-h urinary protein level < 3.5g/d with peak value reduction ≥ 50%, accompanied by improved or normal serum albumin, stable renal function.

SECONDARY OUTCOMES:
Rate of complete remission at 24, 48, 96 weeks | Start of randomization until 96 weeks
  The rate of patients achieve complete remission at 24, 48, or 96 weeks.
Rate of partial remission at 24, 48, 96 weeks | Start of randomization until 96 weeks
  The rate of patients achieve partial remission at 24, 48, or 96 weeks.
Median time to achieve complete remission | Start of randomization until 96 weeks
Median time to achieve partial remission | Start of randomization until 96 weeks
Median time of the first relapse of nephrotic syndrome for patients who achieve complete remission or partial remission | Start of randomization until 96 weeks
Proportion of patients with relapse of nephrotic syndrome | Start of randomization until 96 weeks
Rate of treatment failure at the end of the study | Start of randomization until 96 weeks
  Treatment failure: the efficacy has not reached complete or partial remission
The proportion of reappearance proteinuria (but not reach nephrotic syndrome) for patients with complete response | Start of randomization until 96 weeks
The 24-hour urinary protein level and changes from baseline at 24, 48, 96 weeks | Start of randomization until 96 weeks
The serum albumin level and changes from baseline at 24, 48, 96 weeks | Start of randomization until 96 weeks
Changes of serum creatinine at 24, 48, 96 weeks | Start of randomization until 96 weeks
Changes of blood urea nitrogen at 24, 48, 96 weeks | Start of randomization until 96 weeks
Changes of serum uric acid at 24, 48, 96 weeks | Start of randomization until 96 weeks
Changes of serum blood lipid level at 24, 48, 96 week | Start of randomization until 96 weeks
The level and changes of estimated glomerular filtration rate (eGFR) calculating using the CKD-EPI formula at 24, 48, 96 weeks | Start of randomization until 96 weeks
Percentage of patients who serum creatinine doubled for 12 weeks, progress to end-stage renal disease, or receive renal replacement therapy | Start of randomization until 96 weeks
The number and proportion of patients who died for any reason | Start of randomization until 96 weeks
The level of phospholipase A2 receptor (PLA2R) and changes from baseline at 24, 48, 96 weeks | Start of randomization until 96 weeks
The level and changes of immunoglobulin and complement | Start of randomization until 96 weeks
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | Start of randomization until 96 weeks
Incidence and severity of adverse reactions (ADR), serious adverse reactions (SADR) | Start of randomization until 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, PhD, Principal Investigator — Chinese PLA General Hospital, Beijing, China
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No